CLINICAL TRIAL: NCT01303198
Title: Autoset T Versus CPAP- Ein Titrations- Und Therapievergleich
Brief Title: Autoset T Versus CPAP Therapy, a Comparison of Titration and Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaiserswerther Diakonie (Other)
Collaborators: ResMed Foundation (Other)
Responsible Party: Hartmut Grueger, Kaiserswerther Diakonie
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Kaiserswertherdiakonie
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Sleep Apnea Syndromes
Keywords: CPAP; APAP; sleep apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP (Active Comparator): Use of CPAP as treatment for sleep apnea
  Interventions: Device: APAP - Therapy
- APAP (Active Comparator): Use of APAP as treatment for sleep apnea
  Interventions: Device: APAP - Therapy

INTERVENTIONS:
Device: APAP - Therapy — automatic positive pressure therapy

SUMMARY:
Part 1.Comparison of manual pressure titration in laboratory of sleep disorders with Autoset T APAP device from Resmed. Hypothesis: There is no difference in efficiency between manual and automatical titration.

Part 2. Comparison of CPAP and APAP therapy in the home while 3 month by Questionaire and device data.

Hypothesis: There is a difference in compliance and efficiency between CPAP and APAP mode.

DETAILED DESCRIPTION:
A cross over, simple blind study design has been created for a controlled trial to compare pressure titration and therapy with the Autoset T device.

Part 1: After a baseline polysomnography (PSG) a selected group of patients with obstructive sleep apnea will be titrated in two more nights in a sleep lab under APAP mode and CPAP mode. We compare the sleep quality and the AHI, oxygen saturation, leakage.

Part 2: Over a time range of 12 weeks the patients got two kinds of therapy modes at home: CPAP and APAP (each six weeks. We compare the objective and subjective therapy by compliance, device data, Epworth sleepiness scale, Pittsburgh Sleep Quality Index (PSQI, german version).

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 80 years

Exclusion Criteria:

* pregnancy
* insomnia
* consumption of soporifics
* pulmonal or cardial diseases
* operation advised by ear, nose and throat specialist
* missing linguistic skills in german

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-06; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
AHI- score (apnea- hypopnea- index) | 3 months
  AHI (apnea- hypopnea- index): Number of Apneas and Hypopneas/hour as a function of the type of positive airway pressure supply used- automated (APAP) vs. the standard, manually titrated and fixes continuous (CPAP).

SECONDARY OUTCOMES:
Number of device-using hours | 3 months
  Number of device-using hours as a means to assess patient compliance with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Grueger, Arzt, Principal Investigator — Diakonie Kaiserswerth
Locations (1):
- Florence-Nightingale-Krankenhaus, Düsseldorf, Nordrhein Westphalen, Germany